CLINICAL TRIAL: NCT05078489
Title: Acute Effects of Action Observation on Pain Intensity, Muscle Strength, Tactile Acuity and Pressure Pain Threshold.
Brief Title: Acute Effects of Action Observation on Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Responsible Party: Principal Investigator, Anabela G Silva, Assistant Professor, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-CED/2020
Record Dates: First submitted 2021-10-04; First posted 2021-10-14 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Action-observation arm (Experimental): Participants will be asked to watch videos of neck exercises without performing any exercise. The intervention will take approximately 15 minutes.
  Interventions: Other: Action-observation therapy
- Placebo intervention (Placebo Comparator): Participants will be asked to watch videos of landscapes. The intervention will take approximately 15 minutes.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Action-observation therapy — Action observation therapy involves the observation and perception of human movement performed by others. The observation of actions performed by others activates in the perceiver the same neural structures responsible for the actual execution of those same actions.
  Arms: Action-observation arm
Other: Placebo — Participants will watch a natural landscape without any human.
  Arms: Placebo intervention

SUMMARY:
This study aims to assess the immediate effects of action observation therapy on the cervical muscles' strength, pain intensity, tactile acuity and pain pressure threshold in individuals with chronic nonspecific neck pain.

DETAILED DESCRIPTION:
This study is a randomized controlled trial with two arms: action observation group vs control group. The action observation group will be asked to watch videos of neck exercises with full attention and concentration and not perform any motion or execute any movement during the observation time. The control group will be asked to watch videos of a landscape.

Participants will be assessed at baseline and at post-intervention for muscle strength, pain intensity, pressure pain threshold and tactile acuity.

ELIGIBILITY:
Inclusion Criteria:

* Have nonspecific chronic neck pain, defined as a recurrent or persistent pain that lasts more than 3 months, with no trauma or etiology/diagnosis associated.

Exclusion Criteria:

* Visual and hearing dysfunction not corrected by eyeglasses/contact lenses or a hearing aid;
* Infectious diseases;
* Cervical myelopathy;
* Cervical surgery;
* Cervical fracture or/and subluxation;
* Vestibular pathology;
* Neurological disorder/deficits;
* Rheumatic autoimmune diseases;
* History of cancer;
* Severe cervical trauma.

Ages: 18 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-20 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Pressure pain thresholds | Baseline
  Pressure pain thresholds are the minimum amount of pressure applied with an algometer that is perceived as being painful; is measured in Kgf
Pressure pain thresholds | Post-intervention (within the same session of the baseline assessment but approximately 30 minutes after that).
  Pressure pain thresholds are the minimum amount of pressure applied with an algometer that is perceived as being painful; is measured in Kgf

SECONDARY OUTCOMES:
Pain intensity | Baseline
  Measured with a 100 mm Visual Analogue Scale
Pain intensity | Post-intervention (within the same session of the baseline assessment but approximately 30 minutes after that).
  Measured with a 100 mm Visual Analogue Scale
Tactile acuity | Baseline
  Assessed as the ability of the participant to distinguish two points using a caliper and the measurement units is millimetres.
Tactile acuity | Post-intervention (within the same session of the baseline assessment but approximately 30 minutes after that).
  Assessed as the ability of the participant to distinguish two points using a caliper and the measurement units is millimetres.
Neck flexors strength | Baseline
  A dynamometer will be used against the forehead of the participants to quantify the isometric strength and units of measurement will be Newtons.
Neck flexors strength | Post-intervention (within the same session of the baseline assessment but approximately 30 minutes after that).
  A dynamometer will be used against the forehead of the participants to quantify the isometric strength and units of measurement will be Newtons.
Neck extensors strength | Baseline
  A dynamometer will be used against the posterior part of the head of the participants to quantify the isometric strength and units of measurement will be Newtons.
Neck extensors strength | Post-intervention (within the same session of the baseline assessment but approximately 30 minutes after that).
  A dynamometer will be used against the posterior part of the head of the participants to quantify the isometric strength and units of measurement will be Newtons.
Neck lateral flexors strength | Baseline
  A dynamometer will be used against the lateral aspect of the head of the participants to quantify the isometric strength and units of measurement will be Newtons.
Neck lateral flexors strength | Post-intervention (within the same session of the baseline assessment but approximately 30 minutes after that).
  A dynamometer will be used against the lateral aspect of the head of the participants to quantify the isometric strength and units of measurement will be Newtons.

OTHER OUTCOMES:
Catastrophizing | Baseline
  Measured with the Catastrophizing Scale (range 0-52 and higher values are indicative of higher pain catastrophizing)
Disability | Baseline
  Measured using the Neck Disability Index (Range: 0 - 50 and higher values indicate higher disability)
Fear of movement | Baseline
  Measured with the TAMPA Scale of Kinesiophobia (range: 13-52 and higher values are indicative of higher levels of fear of movement)
Fear-avoidance beliefs | Baseline
  Measured with the Fear-Avoidance Beliefs Questionnaire (range: 0-66 with higher scores indicating higher fear-avoidance beliefs)

CONTACTS AND LOCATIONS:
Overall Officials: Anabela o Silva, Principal Investigator — School of Health Sciences, University of Aveiro
Locations (1):
- School of Health Sciences, University of Aveiro, Aveiro, Portugal

REFERENCES:
- [Derived] Al Shrbaji T, Bou-Assaf M, Andias R, Silva AG. A single session of action observation therapy versus observing a natural landscape in adults with chronic neck pain - a randomized controlled trial. BMC Musculoskelet Disord. 2023 Dec 19;24(1):983. doi: 10.1186/s12891-023-07070-w. PMID 38114952